CLINICAL TRIAL: NCT01507311
Title: Effect of NNC90-1170 on Pulsatile Insulin Secretion in Type 2 Diabetic Patients. A Double-blind, Placebo-controlled, Randomised, Single-dose, Cross-over Trial
Brief Title: Effect of Liraglutide on Pulsatile Insulin Secretion in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1219
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — A single dose injected subcutaneously (under the skin)
  Other Names: NNC 90-1170
  Arms: NNC 90-1170
Drug: placebo — A single dose injected subcutaneously (under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the effect of NNC 90-1170 (liraglutide) on pulsatile insulin secretion and insulin secretion after a standard meal in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes, either newly diagnosed with at least two months of diet treatment, or in current OHA (oral hypoglycaemic agent) treatment with stable dose for at least six months
* BMI (Body Mass Index) between 24 and 35 kg/m^2 (both inclusive)
* Fasting plasma glucose between 6 and 15 mmol/l (both inclusive)
* Anti-GAD (glutamic acid decarboxylase) negative

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Receipt of any investigational drug within three months prior to this trial
* Recurrent severe hypoglycaemia as judged by the investigator
* Cardiac disease or any clinically significant abnormal ECG (electrocardiogram)
* Use of any drug (except oral hypoglycaemic agents (OHAs)) which in the investigator's opinion could interfere
* with the blood glucose level (i.e., insulin, systemic corticosteroids, thiazides)
* Liver or renal disease

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1999-09; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Insulin secretory burst mass

SECONDARY OUTCOMES:
Insulin secretory pulse mass, amplitude, frequency and regularity
Insulin secretion
Glucagon response
Gastric emptying rate
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Juhl CB, Hollingdal M, Sturis J, Jakobsen G, Agerso H, Veldhuis J, Porksen N, Schmitz O. Bedtime administration of NN2211, a long-acting GLP-1 derivative, substantially reduces fasting and postprandial glycemia in type 2 diabetes. Diabetes. 2002 Feb;51(2):424-9. doi: 10.2337/diabetes.51.2.424. PMID 11812750
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com